CLINICAL TRIAL: NCT06052150
Title: Improving Gaps in Periodontal Care in Patients With Cirrhosis Through Interventions
Brief Title: Oral Health In Cirrhosis of the Liver (ORACLE)
Acronym: ORACLE
Status: Recruiting | Type: Observational
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Collaborators: Virginia Commonwealth University (Other); Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: BAJAJ0034
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Cirrhosis; Periodontal Diseases
MeSH Terms: conditions — Fibrosis; Periodontal Diseases | interventions — Diagnosis, Oral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plaque and saliva for microbiota
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cirrhosis: Outpatients with cirrhosis with the following criteria
  Inclusion criteria A. Age>18 years B. Cirrhosis confirmed (liver biopsy, signs of current or prior decompensation, varices in patients with chronic liver disease, nodular liver on imaging, AST>ALT and platelet count >150K in patients with chronic liver disease, ultrasound, or MR elastography suggestive of cirrhosis).
  C. Willing and able to give consent Exclusion criteria A. Unclear diagnosis of cirrhosis B. Unable or unwilling to consent C. Edentulous D. Prior organ transplant E. On anticoagulant therapy
  Interventions: Procedure: Dental exam and periodontal cleaning if needed

INTERVENTIONS:
Procedure: Dental exam and periodontal cleaning if needed — Dental exam and periodontal cleaning if needed

SUMMARY:
The goal of this observational study is to learn about dental evaluation and periodontal cleaning along with scheduled follow -up on the dental health and overall health of patients with cirrhosis and also to determine what barrier(s) if any exist to improve oral health in this population.

DETAILED DESCRIPTION:
Oral health is a major concern for access across the USA. This is especially important in patients with cirrhosis, who have impaired oral and systemic immune responses, microbial alterations in the mouth and saliva, and repeated admissions and medication exposures. In addition, the higher rate of alcohol and smoking in this population exacerbates the impaired oral health. Patients with cirrhosis also have a very high rate of periodontitis, which can lead to systemic inflammation and can lead to poor outcomes. Access to dental care is relatively poor due to financial concerns and lack of dental insurance and currently is only required for liver transplant assessment. Cirrhosis and chronic liver disease is also associated with poor socio-economic status, which worsens the access issues. In addition, low awareness of oral health in cirrhosis from medical practitioners makes it even harder to convince patients of this need for routine dental care. In addition to the lack of access, there is evidence that the oral and subgingival microbiome in cirrhosis can have systemic impacts. Salivary microbiome is altered favorably after rifaximin therapy and after cleaning of teeth by dental professionals in patients with cirrhosis. In NACSELD3 experience, history of periodontitis was independently associated with 3-month hospitalizations (Published in Clinical Gastroenterology and Hepatology). However, if patients are not seen in dental clinics, oral conditions including periodontitis cannot be reliably diagnosed, and treated adequately and appropriately according to diagnosed condition. Therefore, the first step towards diagnosing and treating periodontitis is to provide access to dental care in patients with cirrhosis and then study the impact of potential therapies on outcomes.

Aims:

A. Determine the status of dental care and access in patients with cirrhosis in outpatient settings B. For those who do not have regular dental care, determine reasons why using semi-quantitative questions and also what would motivate them to seek regular dental care.

C. Determine the oral health status, rate and severity of periodontitis for those who agree to get a dental and periodontal examination D. Determine why patients attend/ do not get regular dental care. E. Determine the impact of dental care and presence of periodontitis on outcomes over time

Patients with cirrhosis who are eligible will be approached and informed of this protocol. Semi-quantitative questionnaires will be administered before/after dental care visits.

Their dental visit will consist of comprehensive dental (D0150) and periodontal examination (D0180) and Panoramic radiograph and bitewings if deemed necessary to facilitate dental disease and periodontal diagnoses. Additionally, a head and neck exam, intraoral exam and review of radiographic findings on PANORAX will be performed and any deviations from health will be noted during this initial examination. Dental examination will diagnose dental disease (caries, fractured teeth etc.), endodontic pathology, retained roots and conditions on oral mucosa and tongue. Periodontal examination will include recordings of probing depths, free gingival margin, clinical attachment loss, recession, furcation involvement and mobility of teeth. Based on clinical and radiographic findings, a detailed periodontal diagnosis and treatment recommendations for initial therapy will be performed if desired and further plans will be suggested.

In addition, during the visit salivary samples, and 4 quadrant subgingival plaque specimens will be collected that will be stored in RNALater in a coded manner until microbial analysis is performed. These will be stored in a minus 80-degree freezer.

Another semi-quantitative questionnaire will also be administered by the dental clinic Co-I that will ask the patients why they came for the visit

At the end of the visit for those who scheduled it, a treatment plan will be developed by the co-Is at the VCU School of dentistry clinics. This will be dependent on the patient's oral health including treatment of dental and periodontal disease and any other noted pathologic conditions discovered during initial examination. Treatment for periodontal disease will be offered through VCU's undergraduate and graduate periodontal clinics. In case of dental disease, patients will be offered referral and treatment will be provided in the VCU predoctoral dental clinics for disease control phase of treatment. All treatment plans presented to study subjects will adhere to the standard of care guidelines. The treatment plan and options to complete the treatment(s) will be discussed with the patient. However, the treatments following initial exam will not be covered by the study.

Finally subjects' charts will be followed over 1 year for dental and medical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Cirrhosis confirmed (liver biopsy, signs of current or prior decompensation, varices in patients with chronic liver disease, nodular liver on imaging, AST>ALT and platelet count >150K in patients with chronic liver disease, ultrasound, or MR elastography suggestive of cirrhosis).
* Willing and able to give consent

Exclusion Criteria:

* Unclear diagnosis of cirrhosis
* Unable or unwilling to consent
* Edentulous
* Prior organ transplant
* On anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Access to dental care | at enrollment.
  Barriers towards dental care will be inquired using a semi-quantitative questionnaire Will be a yes or no answer

SECONDARY OUTCOMES:
Previously undiagnosed periodontitis | at the time of dental exam
  Proportion of subjects examined who had periodontitis; Will be a yes or no answer
Proportion with existing dental care | at enrollment
  Proportion of subjects examined who have pre-existing dental care; Will be a yes or no answer
Death | 1 year; Will be a yes or no answer
  Proportion of subjects examined who died during the 1 year follow-up
Transplant | 1 year
  Proportion of subjects examined who received a liver transplant during the 1 year follow-up; Will be a yes or no answer
Hospitalizations | 1 year
  Proportion of subjects who were hospitalized during the 1 year follow-up; Will be a yes or no answer

OTHER OUTCOMES:
Plaque microbiome diversity | at the time of dental exam
  Shannon diversity of plaque bacteria which is a continuous scale
Salivary microbiome diversity | at the time of dental exam
  Shannon diversity of salivary bacteria which is a continuous scale

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No